CLINICAL TRIAL: NCT03955328
Title: Progression of Damage in Ulcerative Colitis
Acronym: PRODUC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: David Garcia Cinca (Other)
Responsible Party: Sponsor-Investigator, David Garcia Cinca, Fundació Clínic per la Recerca Biomèdica, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HCB/2017/0842
Record Dates: First submitted 2019-05-10; First posted 2019-05-20 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Magnetic Resonance Imaging (Experimental): A magnetic resonance imaging is perform to detect permanent anatomical damage.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging — A magnetic resonance imaging is perform to detect permanent anatomical damage.

SUMMARY:
The hypothesis of the study is that in ulcerative colitis repeated flares of inflammatory activity, as well as mechanisms involved in resolution of the inflammatory response, may contribute to accumulation of damage in the colon leading to functional disturbances and symptoms that affect patient's functioning. The primary objective is to determine whether ulcerative colitis induces permanent anatomical damage, by means of magnetic resonance imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes aged >18 years and <72 years.
* Ulcerative colitis diagnosed according to European Crohn's and Colitis Organization guidelines .
* Ulcerative colitis in endoscopic remission as demonstrated by a recto-sigmoidoscopy/colonoscopy (defined as: Mayo Endoscopic Score 0-1; Ulcerative Colitis Endoscopic Index of Severity : bleeding 0, vascular 0-1, erosion/ulcers 0).
* Normal C-reactive protein according local laboratory values.
* Informed consent for participation.
* Understands the language of the provided patient questionnaires.

Exclusion Criteria:

* Pregnant women (or pregnancy suspected).
* Previous colonic surgery.
* Patients receiving corticosteroids or antidiarrheal medications.
* Patients with suspected or confirmed active gastrointestinal infection.
* Patients with a diagnosis of other gastrointestinal disorders that may result in symptoms including, but not limited to, celiac disease, intolerance to disaccharides and pancreatic disorders.
* Diabetes.
* Thyroid disorders.
* Liver disease.
* Any other systemic disease that, according to the investigator's criteria, might influence the variables investigated.
* Patients with history of colonic dysplasia.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-06-15 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-06-15 (Estimated)

PRIMARY OUTCOMES:
Relationship of structural changes in colon morphology and functional changes assessed by MRI with disease duration in UC patients in clinical remission | Baseline
  Explorative structural changes

SECONDARY OUTCOMES:
Patient reported outcomes on IBDQ-32 questionnaire | Baseline
  Inflammatory bowel diseases health-related quality of life index which is a questionnaire of 32 items, score ranges from 32 to 224.
Patient reported outcomes on EQ-5D-5L questionnaire | Baseline
  EQ-5D-5L questionnaire a standardized instrument for measuring generic health status, score ranges from -0.224 to 1.
Patient reported outcomes on Work Productivity and Activity questionnaire | Baseline
  Work Productivity and Activity Impairment questionnaire is a well validated instrument to measure impairments in work and activities. Consists in 6 questions: question1: yes/no, questions 2 to 4: number of hours (count data), question 5: global rating scale, 0-10 (0 = health problems had no effect on my work, 10 = health problems completely prevented me from working), question 6: global rating scale, 0-10 (0 = health problems had no effect on my daily activities, 10 = health problems completely prevented me from doing my daily activities)
Patient reported outcomes on Disability Index questionnaire | Baseline
To identify disease characteristics associated with permanent/accumulated damage disease severity with number of f the hospital admissions | Baseline
To identify disease characteristics associated with permanent/accumulated damage disease severity with dose of corticoesteroids | Baseline
To identify disease characteristics associated with permanent/accumulated damage disease severity with dose of immunosuppressants | Baseline
To identify disease characteristics associated with permanent/accumulated damage disease severity with dose of biologics drugs | Baseline
To identify disease characteristics associated with permanent/accumulated damage with the disease extension at diagnosis and maximal extension of the disease at any time proctitis | Baseline
To identify disease characteristics associated with permanent/accumulated damage with the disease extension at diagnosis and maximal extension of the disease at any time left colitis | Baseline
To identify disease characteristics associated with permanent/accumulated damage with the disease extension at diagnosis and maximal extension of the disease at any time extensive colitis | Baseline
To identify disease characteristics associated with permanent/accumulated damage with the time since the disease diagnosis | Baseline
To identify disease characteristics associated with permanent/accumulated damage related to anorectal function using Cleveland Clinic Incontinence Score | Baseline
  Cleveland Clinic Incontinence Score is a questionnaire that reports the consistency and frequency of depositions is a 5 questions questionnaires with 7 possible answers each question.

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Hospital Galdakao, Galdakao, Bizkaia
  - Hospital Reina Sofía, Córdoba, Cordoba
  - Hospital Puerta de Hierro, Majadahonda, Madrid
  - Hospital Clínic de Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided